CLINICAL TRIAL: NCT01842360
Title: Randomized Double-blind Placebo-controlled Multicenter Clinical Trial of Bacterial Polyvalent Vaccine (BACTEK®), Administered Sublingually in COPD Patients, to Evaluate Efficacy, Safety, and Immunomodulatory Response.
Brief Title: Evaluation of the Efficacy and Safety of MV130 in Chronic Obstructive Pulmonary Disease (COPD)
Acronym: MV130
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Inmunotek S.L. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MV130-SLG-001; 2012-003253-28 (EudraCT Number)
Record Dates: First submitted 2013-04-22; First posted 2013-04-29 (Estimated); Results first posted 2025-10-02 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Chronic Obstructive Pulmonary Disease (COPD)
Keywords: Vaccine; Chronic obstructive pulmonary disease (COPD); Exacerbations; Prevention; Sublingual
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active - MV130 (Experimental): The participants will receive daily dose of MV130 during 12 months sublingually.
  Interventions: Biological: MV130
- Placebo (Placebo Comparator): The participants will receive daily dose of placebo during 12 months sublingually.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Placebo — The participants will receive daily dose of placebo during 12 months sublingually.
  Arms: Placebo
Biological: MV130 — The participants will receive daily dose of MV130 during 12 months sublingually.
  Arms: Active - MV130

SUMMARY:
The goal of this clinical trial is to learn whether the bacterial vaccine MV130 helps reduce the number of exacerbations in adults with moderate to severe COPD. It will also assess the safety and immune effects of MV130. The main questions it aims to answer is: Does MV130 lower the number and severity of COPD flare-ups? Other questions include: Does it reduce the use of healthcare resources and improve quality of life?

Researchers will compare MV130 to a placebo (a similar spray without the active substance; bacterial species) to see how well it works. Participants will use either MV130 or placebo daily under the tongue for 12 months, attend regular clinic visits, and be followed for an additional 6 months to monitor health outcomes and side effects.

DETAILED DESCRIPTION:
This was a randomized, double-blind, placebo-controlled, prospective, parallel, multicenter clinical trial designed to evaluate the efficacy, safety, and immunomodulatory effects of a sublingually administered bacterial polyvalent vaccine (BACTEK®, also known as MV130) in adult participants with moderate to severe Chronic Obstructive Pulmonary Disease (COPD). The study was conducted by Inmunotek, S.L., and included seven sHospitals across Spain. A total of 198 participants were enrolled and randomized equally into two groups to receive either MV130 or placebo over a period of 12 months, followed by a 6-month observation phase, totaling 18 months of participation per participant.

The investigational product, MV130, consisted of a glycerinated suspension containing six inactivated non-lysate bacterial species: Streptococcus pneumoniae, Staphylococcus epidermidis, Staphylococcus aureus, Klebsiella pneumoniae, Moraxella catarrhalis, and Haemophilus influenzae. The product was administered sublingually at a dosage of two sprays (0.2 mL total) per day. The placebo formulation was identical in appearance and composition, excluding the active bacterial components. All study participants received their first dose under supervision at the clinical site and were trained for home administration.

Eligible participants were between 35 and 85 years old, with a diagnosis of moderate or severe COPD according to GOLD guidelines, a history of recurrent exacerbations (≥3 moderate or ≥2 with at least one hospitalization in the past year), and a smoking history of at least 10 pack-years. Subjects were excluded if they had very severe COPD, a history of recent exacerbations or systemic corticosteroid use, concurrent immunodeficiency or serious comorbid conditions, or if they were pregnant, breastfeeding, or unwilling to use contraception during the study.

The primary efficacy endpoint was the total number of COPD exacerbations during the full 18-month period. Secondary endpoints included the severity of exacerbations, time to first exacerbation, healthcare resource usage (hospitalizations, emergency room visits, unscheduled consultations), medication use, health-related quality of life (assessed using the CAT questionnaire), and a pharmacoeconomic evaluation based on healthcare expenditures. In a subset of participants, immunological parameters were also assessed to explore the immunomodulatory response. Safety analysis included all randomized participants.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent.
* Both sexes.
* Age between 35 and 85.
* Must be capable of complying with the dosing regimen.
* Diagnosis of moderate or severe COPD according to GOLD criteria.
* Experienced at least three moderate exacerbations (i.e., those requiring treatment with antibiotics, systemic corticosteroids, or both, as prescribed by their general practitioner or pulmonologist in the standard consultation and/or the Emergency Department of their Clinic) or two exacerbations with at least one requiring hospitalization due to a COPD exacerbation and the other one a moderate exacerbation occurred within the last year.
* Not changed their medication for the maintenance treatment of COPD within the past 6 months.
* Consumption of 10 or more packs of cigarettes/year. Participants may be or not active smokers.
* Live in the Autonomous Community of Madrid throughout the study period.
* Women of childbearing age women of must use an approved contraceptive method and obtain a negative result in the urine pregnancy test performed during the screening visit.

Exclusion Criteria:

* Participants outside allowed age range.
* Participants unable to cooperate and/or have a severe psychiatric disorder.
* Women who are pregnant, breastfeeding, expect to become pregnant during the study (including assisted reproduction), or who refuse to use contraceptives during the study (including barrier methods). Women who become pregnant during the clinical trial will have to discontinue their participation in it.
* Participants who has participated in a study or clinical trial with an investigational product in the last 3 months before inclusion.
* Participants diagnosed with asthma based on the guidelines of the American Thoracic Society and the European Respiratory Society. If the investigators are unable to differentiate between COPD and asthma after applying the criteria listed in the following table, a bronchodilator test with inhaled salbutamol must be performed, excluding those subjects with FEV1 changes >400 ml.
* Participants with a diagnosis other than COPD that causes them to have an unstable condition or a life expectancy <3 years.
* Participants who had an exacerbation within 4 weeks before starting the trial.
* Participants with moderate COPD who required treatment with inhaled corticosteroids in the last 4 weeks.
* Participants with moderate COPD who received systemic corticosteroids (orally, intramuscularly, or intravenously) in the last 4 weeks.
* Participants diagnosed with a Primary or Secondary Immunodeficiency within the 12 months preceding their inclusion in the clinical trial or the trial's baseline visit.
* Participants diagnosed with chronic lymphoproliferative disease.
* Participants diagnosed with chronic infectious disease.
* Participants with chronic heart disease, arrhythmias, or episodes of arrhythmia secondary to the administration of bronchodilators.
* Participants diagnosed with COPD and chronic colonization by Pseudomonas aeruginosa.
* Participants with COPD and bronchiectasis diagnosed by CT imaging before the age of 40.
* Participants diagnosed with very severe COPD according to the GOLD classification.
* Participants requiring home oxygen therapy or non-invasive mechanical ventilation.
* Participants with a history of hypersensitivity to any of the vaccine's components.
* Participants receiving immunosuppressive treatment with: azathioprine, methotrexate, ciclosporin, cyclophosphamide, tacrolimus, antimalarial drugs, or gold salts.
* Participants who have been treated with monoclonal antibodies such as rituximab or TNF-alpha inhibitors in the last 6 months.
* Participants receiving chronic treatment with azithromycin or inhaled antibiotics (tobramycin or colistin).

Ages: 35 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2013-05-06 (Actual); Primary Completion 2019-07-29 (Actual); Study Completion 2023-08-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eduardo Fernández Cruz, MD, PhD, Study Director — Hospital General Universitario Gregorio Marañón; Javier de Miguel Díez, MD, PhD, Principal Investigator — Hospital General Universitario Gregorio Marañón; José Luis Álvarez-Sala, MD, PhD, Principal Investigator — Hospital San Carlos, Madrid; María J Buendía, MD, Principal Investigator — Hospital Universitario Infanta Leonor; Carlos J Álvarez, MD, PhD, Principal Investigator — Hospital Universitario 12 de Octubre; Soledad Alonso, MD, Principal Investigator — Hospital Universitario de Torrejón,Madrid; Francisco García, MD, PhD, Principal Investigator — Hospital Universitario La Paz; Joan Serra, MD, Principal Investigator — Hospital de Universitario Vic
Locations (7):
- Spain (7):
  - Hospital Universitario de Vic, Vic, Barcelona
  - Hospital Universitario de Torrejón, Torrejón de Ardoz, Madrid
  - Hospital General Universitario Gregorio Marañón, Madrid
  - Hospital Universitario Infanta Leonor, Madrid
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario La Paz, Madrid

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- MV130: The participants will receive daily dose of MV130 during 12 months
  MV130: The participants will receive daily dose of MV130 during 12 months
- Placebo: The participants will receive daily dose of placebo during 12 months
  Placebo: The participants will receive daily dose of placebo during 12 months
Period: Overall Study
Arm/Group | MV130 | Placebo
Started | 97 | 101
Completed | 63 | 79
Not Completed | 34 | 22

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MV130 | Placebo | Total
Number analyzed (Participants) | 97 | 101 | 198
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.0 (9.3) | 70.0 (8.9) | 69.0 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 25 | 44
  Male | 78 | 76 | 154
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 97 | 100 | 197
  Unknown or Not Reported | 0 | 0 | 0
Weight [Mean (Standard Deviation); unit: kilograms] | 76.2 (15.6) | 73.5 (15.2) | 74.8 (15.4)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index
  kg/m^2 | 27.8 (4.5) | 27.5 (4.7) | 27.6 (4.6)
FEV1 [Mean (Standard Deviation); unit: liters] — Forced Expiratory Volume in 1 second
  liters | 55.7 (14.5) | 56.9 (14.6) | 56.3 (14.5)
Smoking status [Number; unit: Participants] — current smokers at baseline visit
  Participants | 21 | 22 | 43
CAT [Mean (Standard Deviation); unit: Score] — COPD Assessment Test Score
  Score | 13.9 (6.8) | 13.2 (7.2) | 13.5 (6.2)
VAS [Mean (Standard Deviation); unit: scores on a scale] — Visual Analogue Scale (VAS) at baseline. Minimum score is 0 and maximum is 10; 0 being feeling worst and 10 feeling best.
  scores on a scale | 7.1 (1.6) | 7.0 (1.7) | 7.0 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: Number of COPD Exacerbations.
Description: Comparison in the number of COPD exacerbations in the two study groups in the 18-month study period.
Time Frame: 18 months
Measure: Median (Inter-Quartile Range); unit: number of exacerbations
Arm/Group | Active - MV130 | Placebo
Number analyzed (Participants) | 97 | 101
number of exacerbations | 2.0 [1.0 to 3.0] | 3.0 [1.0 to 5.0]
Statistical Analysis 1: Comparison: Active - MV130 vs Placebo; Test type: Superiority; p < 0.01, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Change in the Rate of COPD Exacerbations.
Description: Incidence is the number of new events per total participants in the sample population.
Time Frame: 18 months
Measure: Number; unit: events per participant-year
Arm/Group | Active - MV130 | Placebo
Number analyzed (Participants) | 97 | 101
events per participant-year | 1.86 | 2.67
Statistical Analysis 1: Comparison: Active - MV130 vs Placebo; Test type: Superiority; p < 0.001, Poisson

3. Secondary Outcome: Change in Severity of COPD Exacerbations.
Description: The severity of exacerbations was to be measured by the consumption of health care resources:
  Emergency Department/Hospitalisation/Intensive Care Unit/Consultations visits, as follows:
  ICU hospitalisation 4 points Hospitalisation 3 points Emergency room visit 2 points Consultation resulting in change in usual treatment 1 point
Time Frame: 18 months
Measure: Median (Inter-Quartile Range); unit: points
Arm/Group | Active - MV130 | Placebo
Number analyzed (Participants) | 97 | 101
points | 1.0 [0.0 to 5.0] | 3.0 [1.0 to 23.0]
Statistical Analysis 1: Comparison: Active - MV130 vs Placebo; The mean of health care consumption was 17.5±34.7 points in the placebo group versus 9.2±27.9 points in the MV130 group; Test type: Superiority; p = 0.0094, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Time Elapsed Between Start of Treatment and First COPD Exacerbation.
Description: For reference, median survival or event-free times are reported with the 95% CI of the median.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: number of months
Arm/Group | Active - MV130 | Placebo
Number analyzed (Participants) | 97 | 101
number of months | 6.35 [4.41 to 9.00] | 4.42 [3.38 to 6.61]
Statistical Analysis 1: Comparison: Active - MV130 vs Placebo; Test type: Superiority; p = 0.3917, Log Rank

5. Secondary Outcome: Use of Drugs (Antibiotics, Corticosteroids, Etc).
Description: The use of drugs will be calculated using the following index:
  * antibiotics: 1 point
  * inhaled corticosteroids: 2 points
  * systemic corticosteroids: 3 points
Time Frame: 18 months
Measure: Median (Inter-Quartile Range); unit: points
Arm/Group | Active - MV130 | Placebo
Number analyzed (Participants) | 97 | 101
points | 24.0 [0.0 to 71.0] | 40.0 [9.0 to 112.0]
Statistical Analysis 1: Comparison: Active - MV130 vs Placebo; As for the previous index the number of days with any of these drugs is used; Test type: Superiority; p = 0.0232, Wilcoxon (Mann-Whitney)

6. Secondary Outcome: Number of Hospitalizations Due to a COPD Exacerbation.
Description: The same patient could have more than one hospitalizations.
Time Frame: 18 months
Measure: Median (Inter-Quartile Range); unit: number of hospitalizations
Arm/Group | Active - MV130 | Placebo
Number analyzed (Participants) | 97 | 101
number of hospitalizations | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 1.0]
Statistical Analysis 1: Comparison: Active - MV130 vs Placebo; Test type: Superiority; p = 0.0319, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Days of Hospitalization Due to a COPD Exacerbation.
Description: Number of days of hospitalization per patient were recorded. The same patient could have more than one hospitalization.
Time Frame: 18 months
Measure: Median (Inter-Quartile Range); unit: number of days
Arm/Group | Active - MV130 | Placebo
Number analyzed (Participants) | 97 | 101
number of days | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 6.0]
Statistical Analysis 1: Comparison: Active - MV130 vs Placebo; Test type: Superiority; p = 0.0264, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Number of Visits to the Emergency Room.
Description: Number of individual visits were recorded per patient. One patient could have multiple visits.
Time Frame: 18 months
Measure: Median (Inter-Quartile Range); unit: number of visits
Arm/Group | Active - MV130 | Placebo
Number analyzed (Participants) | 97 | 101
number of visits | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 1.0]
Statistical Analysis 1: Comparison: Active - MV130 vs Placebo; The mean number of emergency room visits was 0.37 (±1.15) for the MV130 group and 0.87 (±1.61) for the placebo group; Test type: Superiority; p = 0.0037, Wilcoxon (Mann-Whitney)

9. Secondary Outcome: Number of Unscheduled Medical Consultations Due to COPD
Description: Number of consultations per patient. One patient could have multiple consultations.
Time Frame: 18 months.
Measure: Median (Inter-Quartile Range); unit: number of consultations
Arm/Group | Active - MV130 | Placebo
Number analyzed (Participants) | 97 | 101
number of consultations | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
Statistical Analysis 1: Comparison: Active - MV130 vs Placebo; The mean number of medical consultations was 0.08 (±0.31) for the MV130 group and 0.31 (±0.88) for the placebo group; Test type: Superiority; p = 0.1008, Wilcoxon (Mann-Whitney)

10. Secondary Outcome: Health Related Quality of Life.
Description: COPD Assessment Test per patient determined by an adapted version of the specific COPD Assessment Test. Minimum value is 0 (better) and maximum value is 40 (worse). The change between two or more time points is reported. Change between baseline and 18 months in shown.
Time Frame: 18 months
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Active - MV130 | Placebo
Number analyzed (Participants) | 97 | 101
score on a scale | -1.5 [-7.0 to 1.5] | -1.0 [-5.0 to 3.0]
Statistical Analysis 1: Comparison: Active - MV130 vs Placebo; Test type: Superiority; p = 0.0367, t-test, 2 sided

11. Secondary Outcome: Healthcare Resource Utilization During COPD Exacerbations
Description: Healthcare resource utilization was assessed as the sum of:
  * Complementary tests
  * Programmed visits to the specialist
  * Total number of visits to the specialist
  * Non-programmed visits to the specialist
  * ICU hospitalization days
  * Visits to the emergency room
  * Days hospitalized
  * Sum of antibiotics
  * Number of visits to General Practitioner
  * Sum of oral corticosteroids
  * Number of telephone calls to the GP
  * Sum of inhalers
  * Home visits
  * Sum of antipyretics
  Total number of healthcare resources used during COPD exacerbation episodes. Data were summarized per treatment group and reported as total counts and percent differences. No baseline or monetary data were collected
Time Frame: 18 months
Measure: Number; unit: Total number of resource units
Arm/Group | Active - MV130 | Placebo
Number analyzed (Participants) | 97 | 101
Total number of resource units | 5202 | 8231

12. Secondary Outcome: Adverse Events and Overall Tolerability (Adverse Reactions).
Description: Total number of adverse events in Active (MV130) and Placebo groups were compared.
Time Frame: 18 months
Measure: Number; unit: number of events
Arm/Group | Active - MV130 | Placebo
Number analyzed (Participants) | 97 | 101
number of events | 116 | 113
Statistical Analysis 1: Comparison: Active - MV130 vs Placebo; Test type: Superiority; p = 0.3234, Fisher Exact

13. Post Hoc Outcome: Number of Exacerbation-Free Participants During the Follow-up Period (Month 12 to Month 18).
Description: Number of Participants who were free of exacerbation during the 6 month follow-up period were compared between active and placebo groups.
Time Frame: 6 month follow-up period
Measure: Count of Participants; unit: Participants
Arm/Group | Active - MV130 | Placebo
Number analyzed (Participants) | 94 | 97
Participants | 67 | 47
Statistical Analysis 1: Comparison: Active - MV130 vs Placebo; Test type: Superiority; p = 0.001, Log Rank

14. Post Hoc Outcome: Number of Exacerbations, Graded by Exacerbation Severity, at Different Study Time Points.
Description: Cumulated rate of COPD exacerbations per participant, graded by severity, at different time points (change from baseline to 3, 6, 12, and 18 months and follow-up (change from month 12 to 18)).
Time Frame: 3, 6, 12, 18 months and follow-up.
Measure: Median (Inter-Quartile Range); unit: number of exacerbations
Arm/Group | Active - MV130 | Placebo
Number analyzed (Participants) | 97 | 101
number of exacerbations
  Mild exacerbations - 3 months | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Mild exacerbations - 6 months | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Mild exacerbations - 12 months | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Mild exacerbations - 18 months | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Mild exacerbations - Follow up | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Moderate exacerbations - 3 months | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 1.0]
  Moderate exacerbations - 6 months | 0.0 [0.0 to 1.0] | 0.0 [0.0 to 1.0]
  Moderate exacerbations - 12 months | 1.0 [0.0 to 1.0] | 1.0 [0.0 to 3.0]
  Moderate exacerbations - 18 months | 1.0 [0.0 to 2.0] | 1.0 [0.0 to 4.0]
  Moderate exacerbations - Follow up | 0.0 [0.0 to 1.0] | 0.0 [0.0 to 1.0]
  Severe exacerbations - 3 months | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Severe exacerbations - 6 months | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Severe exacerbations - 12 months | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 1.0]
  Severe exacerbations - 18 months | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 1.0]
  Severe exacerbations - Follow up | 0.0 [0.0 to 0.0] | 0.0 [0.0 to 0.0]
  Total - 3 months | 0.0 [0.0 to 1.0] | 0.0 [0.0 to 1.0]
  Total - 6 months | 1.0 [0.0 to 1.0] | 1.0 [0.0 to 2.0]
  Total - 12 months | 1.0 [0.0 to 2.0] | 2.0 [1.0 to 4.0]
  Total - 18 months | 2.0 [1.0 to 3.0] | 3.0 [1.0 to 5.0]
  Total - Follow up | 0.0 [0.0 to 1.0] | 1.0 [0.0 to 1.0]

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, 18 months
Arm/Group | MV130 | Placebo
All-Cause Mortality (participants affected / at risk) | 1/97 | 2/101
Serious Adverse Events (participants affected / at risk) | 9/97 | 12/101
Other Adverse Events (participants affected / at risk) | 26/97 | 13/101
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MV130 (N=97) | Placebo (N=101)
metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Aenocarcinoma pancreas (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Unstable angina (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 1
Surgery (Surgical and medical procedures) | 0 | 1
Petit mal epilepsy (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Haemorrhage intracranial (Nervous system disorders) | 1 | 0
Apendicitis (Gastrointestinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary aspergillosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Mycobacterium avium complex infection (Infections and infestations) | 0 | 1
Cytomegalovirus infection (Infections and infestations) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MV130 (N=97) | Placebo (N=101)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 5 | 8
Urinary tract infection (Renal and urinary disorders) | 8 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-12-29): https://cdn.clinicaltrials.gov/large-docs/60/NCT01842360/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/60/NCT01842360/SAP_001.pdf